CLINICAL TRIAL: NCT05653167
Title: Complex Socio-emotional Learning in VR-based Simulation Training Among Persons With Mental Health and/or Substance Use Disorders"
Brief Title: VR as a Facilitator for Participation in Society Among Persons With MHD/SUD
Acronym: SOPATMEDVR1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 326773VR_WP1
Record Dates: First submitted 2021-10-28; First posted 2022-12-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Substance Use Disorders; Mental Disorder
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is the first part of a larger project called "Virtual Reality (VR) as a facilitator for participation in society among persons with mental health/substance use disorders" in which aims to explore,develop and evaluate a VR-based paradigm that facilitates social participation and promotes social recovery of individuals with mental health and/or substance use disorders (MHD/SUD). The overall project comprises three work packages: an exploration study, a development study, and an evaluation study. This study will make up work package 1. The primary aim of this study (WP1) is to explore facilitators and barriers for participation in society among person with MHD/SUD, and to provide an understanding of mechanisms of social participation and social cohesion among persons with MHD/ SUD that may be affected by VR-based interventions. The investigators will derive a socio-emotional learning domain to facilitate key interpersonal and social processes among persons with MHD/SUD in VR-based interventions. To achieve the purpose of this study, the invistigators conduct 10 indepth interviews with service-user with MHD/SUD, 2 focus group interviews with 14 service-providers and an interview-survey with 100 service users. This gives the investigators the possibility to explore facilitators and barriers for social participation as experienced as by individuals with MHD/SUD and identify key interpersonal and social processes suitable to be addressed by tailored VR based interventions.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* receiving services in the municipality due to mental health and or addiction problems.

Exclusion Criteria:

-visual and hearing impairment, neurological disorders, and mental retardation [score ≤70 on the Test of Intelligence].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises persons with a self reported addiction and mental health disorder who receive services in the municipality. Further, we interview staff (nurses, mental health workers, psycologists, social workers) from the municipal mental health and addiction services.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Practical and social functioning | 2 hours
  measured by the Practical and Social Functioning Scale (PSF)
Social inclusion | 2 hours
  Measured by the Social and Community Opportunities Profile (SCOPE)
Barriers for participation in society | duration of the in-depth interview
  This will be assessed within in-depth interviews
Facilitators for participation in society | duration of the in-depth interview
  This will be assessed within in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lien, MD, Ph.d, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Brumunddal, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT05653167/Prot_000.pdf